CLINICAL TRIAL: NCT00003640
Title: A Feasibility Study of Thorough Transurethral Resection (TURB) and Escalated Dose M-VAC Chemotherapy as Primary Treatment of T2-T3a, N0-Nx, M0 Transitional Cell Carcinoma of the Bladder, With the Intention of Bladder Preservation
Brief Title: Transurethral Resection and Combination Chemotherapy in Treating Patients With Stage II or Stage III Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-30971; EORTC-30971
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Methotrexate; Vinblastine; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: vinblastine sulfate
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combination chemotherapy combined with transurethral resection may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of transurethral resection plus combination chemotherapy in treating patients who have stage II or stage III bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the percentage of patients with transitional cell carcinoma of the bladder who are disease free or who have minimal disease 3 months after thorough transurethral resection (TURB) and escalated dose methotrexate/vinblastine/doxorubicin/cisplatin (M-VAC) chemotherapy. II. Evaluate the combination of thorough TURB and escalated dose M-VAC followed by radiotherapy with respect to bladder preservation for patients who respond to neoadjuvant chemotherapy. III. Evaluate the proportion of patients remaining disease free and not requiring cystectomy at 1 year. IV. Evaluate the feasibility and morbidity of this treatment schedule in multiple institutions applied by urologists of possibly varying endoscopic ability.

OUTLINE: This is a multicenter study. Patients undergo a local transurethral resection. Patients then receive methotrexate IV on day 1, followed by vinblastine IV, doxorubicin IV, and cisplatin IV on day 2. Filgrastim (G-CSF) is administered on days 4-10. Chemotherapy is repeated every 14 days for 3 courses. After the end of chemotherapy, patients undergo another local transurethral resection in order to define response to treatment. Patients with minimal or no disease are treated with radiotherapy. Patients who still have disease undergo a cystectomy. Patients are followed every 3 months for the first 2 years, and then every 6 months until death.

PROJECTED ACCRUAL: A total of 29-73 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Transitional cell carcinoma of the bladder with biopsy proven muscle invasion suitable for resection leaving no residual visible or palpable tumor mass Unifocal No greater than 5 cm Stages II and III (T2-T3a, N0-NX, M0) No prior treatment for bladder cancer other than endoscopic resection, intravesical chemotherapy, or intravesical immunotherapy

PATIENT CHARACTERISTICS: Age: Not specified Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 120,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT normal Renal: GFR at least 50 mL/min Cardiovascular: Normal cardiac function (i.e., no New York Heart Association class II-IV) Other: Normal auditory function No second primary malignant tumor except basal cell carcinoma of the skin Fit for cisplatin containing combination chemotherapy, radical radiotherapy, or cystectomy No active infections Not pregnant or nursing No concurrent illness that significantly affects clinical assessments

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics No prior systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the bladder Surgery: See Disease Characteristics No prior partial cystectomy Prior transurethral resection of the bladder allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 1998-09; Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cora N. Sternberg, MD, FACP, Study Chair — Istituto Scientifico H. San Raffaele
Locations (1):
- San Raffaele Hospital, Rome, Italy